CLINICAL TRIAL: NCT06422832
Title: Remote Monitoring To Identify Worsening Heart Failure: The REMOTI-HF Randomized Clinical Trial
Brief Title: Remote Monitoring To Identify Worsening Heart Failure The REMOTI-HF Randomized Clinical Trial
Acronym: REMOTI-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Unidade Local de Saúde de Coimbra, EPE (Other)
Responsible Party: Principal Investigator, Goncalo Terleira Batista, Cardiology Resident, Unidade Local de Saúde de Coimbra, EPE
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: RHF230808
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Heart Failure; Arrythmia
Keywords: Heart Failure; Remote Monitoring; ICD; CRT
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Patients will not know whether the algorithms was activated or not at the beginning of the study. However, if a contact with the patient is made due to the algorithm, the patient will then understand they are not on the control group.
  The person responsible for contacts will also know if an individual patient is on the control or intervention group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interventional group (Experimental): In this group the respective algorithm will be activated and alerts will be sent according to its design
  Interventions: Other: HeartLogic or TriageHF Algorithms for implantable devices
- Control Group (No Intervention): The algorithm will not be activated and follow-up will continue as if the patient was not included in the study.

INTERVENTIONS:
Other: HeartLogic or TriageHF Algorithms for implantable devices — Activation of the HeartLogic and TriageHF algorithms for implantable devices and correctly act according to its design
  Arms: Interventional group

SUMMARY:
Heart failure, characterized by high mortality and morbidity rates, frequent hospital admissions, and prolonged stays in cardiology wards, significantly impacts patients' quality of life.

The REMOTI-HF is a single-center randomized controlled trial designed to assess the impact of remote monitoring, utilizing the HeartLogic and TriageHF algorithms, in patients with heart failure with implantable cardioverter defibrillator or cardiac resynchronization therapy. The primary endpoints include mortality, hospital admissions related to heart failure, and visits for worsening heart failure.

Moreover, we will explore the full capabilities of these algorithms, by analysing the association of physical activity, measured by the devices, with the same key outcomes. Additionally, the research will explore the relationship between the absolute values provided by the algorithms and NT-proBNP values.

DETAILED DESCRIPTION:
Patients will be randomized into two arms: one with the activation of the algorithm and the other with no active algorithm. The algorithm is programmed to alert our team upon detecting a patient at risk of worsening heart failure. When an alarm is triggered, the patient will receive a telephone call from the investigation team. Subsequently, the patient may be scheduled for a hospital visit, or ambulatory medication adjustments can be made.

For patients in whom the algorithm is deactivated, no such alarm mechanism will be in place.

Patients in both arms will undergo comparison based on relevant heart failure events, defined as follows:

* All-Cause Mortality
* Hospital Admission for Heart Failure
* Hospital Visit for Worsening Heart Failure
* Ventricular Arrhythmias
* Atrial Arrhythmias

Additionally, the study will explore the association between physical activity measured by the devices and these specified events.

In addition to evaluating patient outcomes, a correlation analysis will be conducted to examine the relationship between the absolute value provided by the algorithm and absolute NT-proBNP values. This analysis aims to assess the concordance and potential predictive value of the algorithm's output with established biomarkers, specifically NT-proBNP, in the context of heart failure progression and severity (if possible).

ELIGIBILITY:
Inclusion Criteria:

* Possession of an implantable cardioverter defibrillator (ICD) or cardiac resynchronization therapy (CRT) device that is compatible with the HeartLogic or TriageHF algorithms.
* Left ventricular ejection fraction at the time of device implantation must be equal to or less than 35%.

Exclusion Criteria:

* Younger than 18 years old or older than 85 years old.
* Unable to be contacted when out of the hospital.
* Presence of severe cognitive impairment.
* Currently on the heart transplant waiting list

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Primary Composite Outcome | 2 years
  All-cause mortality, Hospital Admission for Heart Failure, Ventricular Arrhythmias and Worsening Heart Failure as defined in the secondary outcome area.

SECONDARY OUTCOMES:
All-cause mortality | 2 years
  All-cause mortality
Hospital admission for Heart Failure | 2 years
  Patient admission to the hospital with symptoms or signs of congestive heart failure, needing intravenous drugs for symptom relief, ultrafiltration therapy, or other parenteral therapy
Worsening Heart failure | 2 eras
  Unscheduled hospital visit (to the emergency department or unscheduled consultation) due to signs or symptoms of heart failure, where intravenous diuretics were administered or ambulatory diuretic dosage was increased.
Ventricular Arrhythmias | 2 years
  Detection of any ventricular arrhythmia through hospital visit, appropriate device therapy or device detection
Atrial Arrhytmias | 2 years
  Occurrence of any atrial arrhythmia prompting medical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Gonçalo Batista, MD, Principal Investigator — ULS Coimbra

IPD SHARING:
Plan to Share IPD: No